CLINICAL TRIAL: NCT07331727
Title: Efficacy of Dapagliflozin on Catheter Ablation Outcomes in Persistent Atrial Fibrillation Patients With Increased Epicardial Adipose Tissue
Brief Title: Epicardial Adipose Tissue-Targeted DApagliflozin for Reducing Electrical Remodeling in Atrial Fibrillation
Acronym: EAT-DARE-AF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Xu Liu, professor, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EAT-DARE-AF
Record Dates: First submitted 2025-12-29; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Atrial Fibrillation (AF)
Keywords: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — dapagliflozin; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin (Experimental): Dapagliflozin 10 mg per day for 3 months after initial catheter ablation
  Interventions: Drug: Dapagliflozin (10Mg Tab) along with standard medical therapy
- Control (No Intervention)

INTERVENTIONS:
Drug: Dapagliflozin (10Mg Tab) along with standard medical therapy — Dapagliflozin 10 mg per day for 3 months after initial catheter ablation
  Arms: Dapagliflozin

SUMMARY:
Persistent atrial fibrillation (PeAF) is associated with a high risk of recurrence following catheter ablation despite advances in ablation technology and strategies. Beyond electrophysiological mechanisms, increasing evidence suggests that atrial structural and inflammatory remodeling plays a pivotal role in the initiation and maintenance of AF, particularly in persistent forms.

Epicardial adipose tissue (EAT) is a metabolically active visceral fat depot located between the myocardium and visceral pericardium. EAT shares a common microcirculation with the underlying atrial myocardium and exerts paracrine and vasocrine effects through the secretion of pro-inflammatory cytokines, adipokines, and profibrotic mediators. Increased EAT volume or thickness has been consistently associated with AF burden, atrial fibrosis, left atrial enlargement, and a higher risk of AF recurrence after catheter ablation.

Sodium-glucose cotransporter 2 inhibitors (SGLT2i) have demonstrated pleiotropic cardiovascular benefits beyond glucose lowering, including reduction in visceral adiposity, attenuation of systemic and local inflammation, and favorable effects on cardiac remodeling. Observational studies and randomized trials in patients with diabetes or heart failure suggest that SGLT2i therapy reduces incident AF and AF recurrence after ablation. However, the effect of SGLT2i in non-diabetic, non-heart failure patients-particularly those with increased EAT as a distinct pathophysiological substrate-remains unclear.This trial is designed to evaluate whether dapagliflozin, administered peri-ablation, can reduce atrial arrhythmia recurrence in PeAF patients with increased EAT but without class I indications for SGLT2i. This targeted approach aims to provide mechanistic and clinical evidence supporting metabolic-inflammatory modulation as an adjunctive strategy to catheter ablation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years;

Diagnosis of persistent atrial fibrillation (continuous AF >7 days and ≤5 years);

Planned first-time catheter ablation for AF;

No class I indications for dapagliflozin, defined as:

No diabetes mellitus;

No history of heart failure (HFrEF, HFmrEF, or HFpEF);

No chronic kidney disease (eGFR ≥60 mL/min/1.73 m²);

Evidence of increased epicardial adipose tissue on cardiac CT or cardiac MRI, defined according to pre-specified imaging thresholds;

Ability to provide written informed consent.

Exclusion Criteria:

* Duration of persistent AF >5 years;

Left atrial anteroposterior diameter >50 mm on transthoracic echocardiography;

Prior AF catheter ablation or surgical ablation;

Current or recent (within 3 months) use of any SGLT2 inhibitor;

Severe structural heart disease (e.g., hypertrophic cardiomyopathy, rheumatic valvular disease, dilated cardiomyopathy);

Contraindications to catheter ablation (e.g., left atrial thrombus, active infection);

Estimated glomerular filtration rate <60 mL/min/1.73 m²;

Type 1 diabetes or history of diabetic ketoacidosis;

Pregnancy or breastfeeding;

Any condition deemed by investigators to make study participation inappropriate.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Atrial fibrillation burden at 3 months after ablation | 3 months
  Atrial fibrillation burden is defined as the percent of time spent in atrial tachyarrhythmia (atrial fibrillation, atrial flutter, or atrial tachycardia) episodes detected by 7-day single-lead ECG patches at 3 months after ablation.

SECONDARY OUTCOMES:
Atrial fibrillation recurrence during 3 months after ablation | 3 months
  Atrial fibrillation recurrence is defined as the first recurrence of any atrial tachyarrhythmia (atrial fibrillation, atrial flutter, or atrial tachycardia) lasting 30 seconds or longer detected by ECG during 3 months after ablation.
Changes of quality of life at 3 months | 3 months
  Changes of quality of life from baseline to 3 months after ablation evaluated by the Atrial Fibrillation Effect on Quality of Life (AFEQT) questionnaire.
Atrial fibrillation recurrence during 1 year after ablation | 1 year
  Atrial fibrillation recurrence is defined as the first recurrence of any atrial tachyarrhythmia (atrial fibrillation, atrial flutter, or atrial tachycardia) lasting 30 seconds or longer detected by ECG during 1 year after ablation.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, China